CLINICAL TRIAL: NCT04639427
Title: Benefits of Using a Transparent Visor to Replace the Face Mask in Speech Therapy Rehabilitation of Oral-Linguo-Facial Praxies in the Context of COVID-19: a Series of Cases
Acronym: Co-VIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200876; IDRCB (Registry Identifier: 2020-A01628-31)
Record Dates: First submitted 2020-11-19; First posted 2020-11-20 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Oral-Linguo-Facial Praxies; Covid19
Keywords: Oral-Linguo-Facial praxies; Covid19; speech therapy rehabilitation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to compare the effectiveness of the use of a transparent covering visor with that of the face mask, with or without the use of video sequences, for speech therapy rehabilitation of oral-linguo-facial praxies in the context of the COVID 19 epidemic.

DETAILED DESCRIPTION:
Statistic analysis: single case experimental design (SCED) method.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 18 years;
* Hospitalization for more than 2 weeks prior to enrollment in the adult post intensive care rehabilitation care unit (PICRU) of Raymond Poincaré hospital in Garches;
* With oral-linguo-facial praxis disorders whatever the cause;
* Has been informed and not in opposition to participation of the study.

Exclusion Criteria:

* Patient with fever or any suspect symptom of a SARS-CoV2 infection;
* Planned discharge of hospital in 2 weeks;
* Patient with cognitive, phasic or vigilance disorders preventing to understand the study;
* Under guardianship or curator;
* Patient Under french AME scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4 patients hospitalized in the adult neurological Post Intensive Care Rehabilitation Unit (PICRU - SRPR) of Raymond Poincaré hospital.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Oral-Linguo-Facial Motricity Test | throughtout of the study, an average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julie PAQUEREAU, MD, Principal Investigator — Unité de Soins de Rééducation Post Réanimation, Service de Médecine Physique et de Réadaptation, Hôpital Raymond Poincaré, APHP
Locations (1):
- Unité de Soins de Rééducation Post Réanimation, Service de Médecine Physique et de Réadaptation, Hôpital Raymond Poincaré, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No